CLINICAL TRIAL: NCT03834909
Title: Correcting Pre-Exposure Prophylaxis (PrEP) Dosing and Adherence Benchmarks in Pregnancy to Optimize HIV Prevention (PrEP-P): A Randomized Comparative Pharmacokinetic Trial
Brief Title: Pre-Exposure Prophylaxis Dosing in Pregnancy to Optimize HIV Prevention (PREP-P)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was not funded
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Record Dates: First submitted 2019-02-06; First posted 2019-02-08 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2021-03

CONDITIONS: Pregnancy; HIV-1-infection
Keywords: HIV Prevention; Healthy Volunteer
MeSH Terms: interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Tenofovir; Emtricitabine

STUDY DESIGN:
Intervention Model Description: The investigators will randomly allocate participants in a 1:1 ratio to two parallel study arms (based on a computer generated randomization scheme).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard Dose Truvada® (Active Comparator): Standard Dose Truvada® - Tenofovir disoproxil fumarate (TDF) 300 mg/Emtricitabine (FTC) 200 mg fixed dose combination (Truvada®), one tablet each day
  Interventions: Drug: Standard dose Truvada®
- Pregnancy-Adjusted Truvada® (Experimental): Pregnancy-Adjusted dose Truvada® - Tenofovir disoproxil fumarate (TDF) 300 mg/Emtricitabine (FTC) 200 mg fixed dose combination (Truvada®), two tablets each day
  Interventions: Drug: Pregnancy-adjusted dose Truvada®

INTERVENTIONS:
Drug: Standard dose Truvada® — TDF/FTC fixed dose combination, 300 mg TDF/200 mg FTC, one tablet each day
  Other Names: Tenofovir Disoproxil Fumarate/Emtricitabine; TDF/FTC
  Arms: Standard Dose Truvada®
Drug: Pregnancy-adjusted dose Truvada® — TDF/FTC fixed dose combination, 300 mg TDF/200 mg FTC, two tablets each day
  Other Names: Tenofovir Disoproxil Fumarate/Emtricitabine; TDF/FTC
  Arms: Pregnancy-Adjusted Truvada®

SUMMARY:
This trial is a prospective, multi-center, randomized comparison study of 2 Pre-Exposure Prophylaxis (PrEP) pharmacokinetic (PK) dosing regimens from 1st trimester through 12 weeks following delivery (postpartum) to achieve study objectives which include PK, safety monitoring for maternal and fetal/infant safety signals, and adherence.

DETAILED DESCRIPTION:
Study participants will be randomized to one of two parallel study arms, involving dosing of tenofovir disoproxil sodium/emtricitabine (TDF/FTC). The investigators will be recruiting and enrolling in the late 1st (preferred) and 2nd trimesters of pregnancy to capture the changes in kidney function and blood flow through the kidneys that appear to start in the late 1st trimester and are most significant in the 2nd and 3rd trimesters of pregnancy. Given the unknown time frame for the return to pre-pregnancy physiologic state and the increased risk of HIV acquisition postpartum, participants will be continued on study dose PrEP until after participants' 1-3 week postpartum visit, after which all participants will be dispensed standard dose PrEP. A 6-12 week postpartum study visit will also be performed to evaluate the timing of return to non-pregnant plasma drug levels during the postpartum period.

PK Sampling. Primary PK data will be derived from up to 7 study visits with PK sampling, including two PK visits in each trimester and postpartum. All PK visits sample blood before an observed PrEP dose. .

Safety Sampling. Maternal safety assessments will continue until 6 months postpartum. Fetal evaluation includes non-invasive limited ultrasound (US) and biophysical profiles (BPP) at study visits and 2nd and 3rd trimester interval growth US, and chart review of all before birth assessments. At birth, the investigators will obtain cord blood plasma to assess for mitochondrial function. Infant safety assessments will continue until 1 year of life. Infants will undergo swaddled Dual-energy X-ray absorptiometry (DXA) scans (without sedation) at 3-6, 24-28, and 50-54 weeks of age. The investigators will assess kidney function by blood sample at 3-6 weeks of life and repeated at 24-28 weeks.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* Able to speak English, French, or Spanish
* Able and willing to provide written informed consent
* Viable first (preferable) or second trimester intrauterine pregnancy
* Creatinine clearance >70 ml/min
* Negative HIV test and no signs/symptoms of acute HIV infection,
* Documented negative hepatitis B virus status.

Exclusion Criteria:

* HIV positive at any time in the study. All neonates of mothers participating in the trial will be recruited, regardless of gestational age at delivery or congenital anomalies/comorbidities.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Must have documented evidence of pregnancy
Enrollment: 0 (Actual)
Dates: Start 2022-04 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Plasma Tenofovir (TFV) Concentration | 36 weeks
  Plasma Tenofovir (TFV) Concentration in nanograms per milliliter (ng/mL)
Plasma Emtricitabine (FTC) Concentration | 36 weeks
  Plasma Emtricitabine (FTC) Concentration in nanograms per milliliter (ng/mL)
Peripheral Blood Mononuclear Cell (PBMC) TFV-Diphosphate (TFV-DP)Concentration | 36 weeks
  PBMC TFV-DP concentration in femtomoles/million cells (fmol/10E6 cells)
Peripheral Blood Mononuclear Cell (PBMC) FTC-Triphosphate (FTC-TP)Concentration | 36 weeks
  PBMC TFV-DP concentration in femtomoles/million cells (fmol/10E6 cells)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Hendrix, MD, Principal Investigator — Johns Hopkins University

IPD SHARING:
Plan to Share IPD: No